CLINICAL TRIAL: NCT01916538
Title: Anorexia Nervosa Genetics Initiative
Acronym: ANGI
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 13-0081
Record Dates: First submitted 2013-07-23; First posted 2013-08-05 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-10

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; genetics; gene; eating disorder
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The blood sample participants provide will be used to identify biological characteristics and other biological "markers." Some analyses will include genetic analyses which are measured using DNA and can look at places in DNA, and others can analyze most of the genome. Other analyses measure a large number of proteins. Still others assess the messenger substance (called RNA) that transfers information from DNA to protein. Investigators plan to store the blood specimens and data indefinitely.
  Investigators will be collecting DNA to permit immediate and future genetic analyses and analyses of immune, endocrine, and proteins. All blood will be biobanked indefinitely to allow for assays that may become available in the future analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Individuals with a current or past diagnosis of anorexia nervosa
- Controls: Individuals who have never been diagnosed with an eating disorder

SUMMARY:
The Anorexia Nervosa Genetics Initiative (ANGI) is the largest and most rigorous genetic investigation of eating disorders ever conducted. Researchers in the United States, Sweden, Australia, and Denmark will collect clinical information and blood samples from over 13,000 individuals with anorexia nervosa and individuals without an eating disorder.

ANGI represents a global effort to detect genetic variation that contributes to this potentially life-threatening illness. The goal of the research study is to transform knowledge about the causes of eating disorders to work toward greater understanding and ultimately a cure.

If you have suffered from anorexia nervosa at any point in your life, you can help us achieve this goal. Your contribution would include a brief questionnaire and a blood sample. If you have never had anorexia nervosa, but still want to contribute, we invite your participation as well.

DETAILED DESCRIPTION:
Participation in this genetics study requires participants to answer some questions online, about eating behaviors (about 15-30 minutes) and to provide a single blood sample that should take only a few minutes.

To obtain the blood sample, investigators will mail you a kit which participants would take to their primary care provider or your local laboratory to have them draw a small sample of blood (about 40 mL, which is less than three tablespoons). The study is also working with a mobile phlebotomy company that can come to your home or location of your choice to draw your blood and ship it at no cost to you. Once the sample is drawn, participants or the mobile phlebotomist will place it in a box and contact FedEx for pick up. There is no cost for the FedEx shipment. Participants will also fill out the reimbursement form and send it and the receipt to our office. Investigators will reimburse participants for the cost of the blood draw. The samples will be studied directly or reprogrammed prior to further study.

ELIGIBILITY:
Inclusion Criteria:

* Lifetime history of anorexia nervosa (cases)

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a lifetime diagnosis of anorexia nervosa
Sampling Method: Non-Probability Sample
Enrollment: 22445 (Actual)
Dates: Start 2013-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Genetic differences | Baseline
  Genetic variation between two groups of people: 1) people with a history of anorexia nervosa and 2) people who have never had an eating disorder will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Bulik, PhD, Principal Investigator — University of North Carolina; Patrick Sullivan, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Thornton LM, Munn-Chernoff MA, Baker JH, Jureus A, Parker R, Henders AK, Larsen JT, Petersen L, Watson HJ, Yilmaz Z, Kirk KM, Gordon S, Leppa VM, Martin FC, Whiteman DC, Olsen CM, Werge TM, Pedersen NL, Kaye W, Bergen AW, Halmi KA, Strober M, Kaplan AS, Woodside DB, Mitchell J, Johnson CL, Brandt H, Crawford S, Horwood LJ, Boden JM, Pearson JF, Duncan LE, Grove J, Mattheisen M, Jordan J, Kennedy MA, Birgegard A, Lichtenstein P, Norring C, Wade TD, Montgomery GW, Martin NG, Landen M, Mortensen PB, Sullivan PF, Bulik CM. The Anorexia Nervosa Genetics Initiative (ANGI): Overview and methods. Contemp Clin Trials. 2018 Nov;74:61-69. doi: 10.1016/j.cct.2018.09.015. Epub 2018 Oct 1. PMID 30287268
- See also: Research study website — http://www.unceatingdisorders.org/angi